CLINICAL TRIAL: NCT01922037
Title: A Prospective Observational Study to Evaluate Predictors of Clinical Effectiveness in Response to Omalizumab
Brief Title: A Study in Participants With Asthma Initiating Treatment With Omalizumab (Xolair)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28528
Record Dates: First submitted 2013-07-12; First posted 2013-08-14 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

ARMS (1):
- Participants With Allergic Asthma (Experimental): Participants with allergic asthma, who have decided to initiate treatment with omalizumab will be observed until a maximum follow-up of 12 months, death, withdrawal of consent, loss to follow-up, or study closure, whichever occurs first.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Participants will receive omalizumab for up to 12 months per investigator standard of care and clinical practice.
  Other Names: Xolair

SUMMARY:
This multicenter, prospective study will evaluate the baseline participant characteristics (including biomarkers) associated with a variety of individual and composite clinical outcomes in participants with moderate to severe asthma initiating treatment with omalizumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants identified by the investigator as a candidate for treatment for asthma with omalizumab
* Confirmation of access to omalizumab through insurance or other source of funding

Exclusion Criteria:

* Enrollment in any other concurrent clinical trial or observational study
* Participants for whom omalizumab treatment is contraindicated
* Participants who had a prior allergic reaction to omalizumab or its excipients
* Participants treated with omalizumab within the previous year
* Participants who received an experimental drug as part of another study within 3 months of enrollment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (145):
- United States (145):
  - Alabama Allergy & Asthma, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Huntsville Lung Associates PC, Huntsville, Alabama
  - San Tan Allergy & Asthma, Gilbert, Arizona
  - Dedicated Clinical Research, Goodyear, Arizona
  - Allergy Associates of Tucson, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Little Rock Allergy & Asthma; Clinical Research Center, Little Rock, Arkansas
  - Stuart Epstein MD - PP, Beverly Hills, California
  - West Coast Clinical Trials Global, LLC, Costa Mesa, California
  - Peninsula Allergy Associates, Daly City, California
  - Allianz Medical and Research Center, Fountain Valley, California
  - William Ebbeling MD - PP, Fresno, California
  - Gettysburg Medical Clinic, Fresno, California
  - Allergy & Asthma Inst Valley, Granada Hills, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Allergy Asthma Care Ctr, Inc., Los Angeles, California
  - Southern California Research Center, Mission Viejo, California
  - North Bay Allergy & Asthma; Medical Assoc, Napa, California
  - Choc Psf, Amc, Orange, California
  - Clinical Trials of Orange County, Orange, California
  - California Allergy & Asthma Medical Group, Inc., Palmdale, California
  - Joann Blessing-Moore MD - PP, Palo Alto, California
  - TPMG - Rancho Cordova, Rancho Cordova, California
  - Redding Allergy & Asthma Care, Redding, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Capital Allergy Resp Dis Ctr, Sacramento, California
  - Central Coast Allergy and Asthma, Salinas, California
  - Allergy Assoc Medical Group, San Diego, California
  - Kaiser Permanente - San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Asthma & Allergy Clinic, San Francisco, California
  - The Allergy and Asthma Clinic, San Mateo, California
  - Allergy & Asthma Medical Group; Clinical Research Division, Walnut Creek, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Christopher C Randolph MD - PP, Waterbury, Connecticut
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - St. Francis Sleep; Allergy & Lung Institute, Clearwater, Florida
  - AAADRS; Clinical Research Center, Coral Gables, Florida
  - Allergy Asthma & Immun Center, Leesburg, Florida
  - Florida Ctr-Allergy & Asthma, Miami, Florida
  - FL Ctr Allergy & Asthma Res, Miami, Florida
  - Allergy & Asthma Care of FL; Clinical Research, Ocala, Florida
  - Central Florida Pulmonary Grou, Orlando, Florida
  - Allergy Asthma & Sinus Center, Palm Beach Gardens, Florida
  - Gulf Coast Allergy Center, P.A., Port Charlotte, Florida
  - USF Asthma Allergy & Immun; Clinical Research, Tampa, Florida
  - Georgia Pollens, Albany, Georgia
  - Brookstone Clinical Res Ctr, Columbus, Georgia
  - Allergy & Asthma Care Center, Gainesville, Georgia
  - Aeroallergy Research Labs, Savannah, Georgia
  - Asthma & Allergy of Idaho, Twin Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Chest Medicine Consultants, Chicago, Illinois
  - Allergy & Asthma Care LTD, Glen Carbon, Illinois
  - Sneeze Wheeze and Itch Associates LLC, Normal, Illinois
  - Allergy Asthma Care, Crown Point, Indiana
  - The Allergy and Asthma Center, Fort Wayne, Indiana
  - Clinical Research Center of Indiana, Indianapolis, Indiana
  - University of Kansas Med Ctr; Int med/Allgy/Immun/Rheum, Kansas City, Kansas
  - Kansas City Allergy And Asthma Assoc., Overland Park, Kansas
  - Abraham Research PLLC, Florence, Kentucky
  - Allergy & Asth Phys of Cent KY, Lexington, Kentucky
  - Dr. Paul Shapero, Bangor, Maine
  - Chesapeake Clinical Research Inc - CRN, Baltimore, Maryland
  - Glenn M. Silber, M.D., P.A, Ellicott City, Maryland
  - Family Allergy & Asthma, Gaithersburg, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Center for Clinical Research., Brockton, Massachusetts
  - Allergy Arth Fam Treatment Ctr, Gardner, Massachusetts
  - Infinity Medical Research Inc, North Dartmouth, Massachusetts
  - McGovern & Baja Allergy Assoc, Springfield, Massachusetts
  - Asthma & Allergy Inst of MI, Clinton Township, Michigan
  - Asthma Allergy Ctr of SW MI, Portage, Michigan
  - Clinical Research Inst, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington Univ. School of Med, St Louis, Missouri
  - Impact Clinical Trials, Las Vegas, Nevada
  - Ocean Allergy & Resp Res Ctr, Brick, New Jersey
  - Adult Ped Aller Central Jersey, Edison, New Jersey
  - Center for Asthma and Allergy, Highland Park, New Jersey
  - Atlantic Allergy Asthma Immunology Associates, Ocean City, New Jersey
  - Allergy Treatment Center of New Jersey, Piscataway, New Jersey
  - Pulmonary and Allergy Associates, Summit, New Jersey
  - Allergy Consultants, PA, Verona, New Jersey
  - SUNY Downstate Medical Center., Brooklyn, New York
  - Boris Sagalovich MD - PC, Brooklyn, New York
  - Island Medical Research Pc, Commack, New York
  - North Shore Medical Arts, LLP, Great Neck, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Winthrop Univ Hospital, Mineola, New York
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Parikh Institute for Research LLC, New York, New York
  - Albert P Hirdt DO - PP, Newburgh, New York
  - Olean Medical Group, Olean, New York
  - University of Rochester, Rochester, New York
  - Advanced Allergy & Asthma PLLC, Rockville Centre, New York
  - Urban Health Plan, Inc., The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Alan Kaufman MD - PP, The Bronx, New York
  - Allergy Partners of Western NC, Asheville, North Carolina
  - Allergy & Asthma Centre of Dayton, Centerville, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Santiago Reyes MD-Private Prac, Oklahoma City, Oklahoma
  - Vital Prospects Clin Res Pc, Tulsa, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Central PA Asth & Allergy Care; Research Division, Altoona, Pennsylvania
  - Allergy and Asthmas; Specialists of Harrisburg, Harrisburg, Pennsylvania
  - Penn State Hershey Medical Group, Hershey, Pennsylvania
  - Inst for Resp & Sleep Med PC, Langhorne, Pennsylvania
  - Allergy and Asthma Research of NJ, lnc, Philadelphia, Pennsylvania
  - Allergy & Clinical Immun Assoc, Pittsburgh, Pennsylvania
  - South Hills Pulmonary Assoc, Pittsburgh, Pennsylvania
  - Respiratory Specialists, Reading, Pennsylvania
  - Nat'l Aller Asth-Charleston, Charleston, South Carolina
  - ADAC Research PA, Greenville, South Carolina
  - Upstate Pharma Research, Simpsonville, South Carolina
  - East Tennessee Center for Clinical Research, Knoxville, Tennessee
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt Medical University, Nashville, Tennessee
  - Greater Austin Allergy Asthma and Immunology, Austin, Texas
  - Elliot J. Ginchansky, MD, PA, Dallas, Texas
  - Allergy Asthma Research Assoc, Dallas, Texas
  - University of Texas Medical Branch;Division of APICS, Galveston, Texas
  - Allergy Asthma & Immun Assoc, Garland, Texas
  - Live Oak Allergy & Asthma Clinic, San Antonio, Texas
  - Allergy & Asthma Res Ctr PA, San Antonio, Texas
  - Sugar Land Allerg Asthma Immun, Sugar Land, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Allergy Associates of Utah, Murray, Utah
  - Bridgerland Clinical Research, North Logan, Utah
  - Pulmonary Research of Albingdon, Abingdon, Virginia
  - O & O Alpan, LLC, Fairfax, Virginia
  - Clinical Research Partners, LLC, Henrico, Virginia
  - Allergy Asthma & Sinus Center, Leesburg, Virginia
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
  - Bellingham Asthma, Allergy & Immunology, Bellingham, Washington
  - ASTHMA, Inc, Seattle, Washington
  - Pulmonary & Sleep Research, Spokane, Washington
  - Northwest Asthma Allergy Center, Vancouver, Washington
  - Allergy Asthma & Sinus Center, Greenfield, Wisconsin
  - Dean Clinic, Madison, Wisconsin
  - University of Wisconsin;Allergy & Asthma Clinical Research, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Fiocchi A, Chinthrajah RS, Ansotegui IJ, Sriaroon P, Mustafa SS, Raut P, Cameron B, Gupta S, Fleischer DM. Does Comorbid Food Allergy Affect Response to Omalizumab in Patients with Asthma? J Asthma Allergy. 2024 Sep 17;17:889-900. doi: 10.2147/JAA.S475517. eCollection 2024. PMID 39309477
- [Derived] Chase NM, Littlejohn M, Holweg CTJ, Millette LA, Seetasith A, Steinke JW, Trzaskoma BL, Hanania NA, Casale TB. Effectiveness of omalizumab across different dosing regimens in patients with moderate-to-severe allergic asthma. Respir Med. 2024 Mar;223:107537. doi: 10.1016/j.rmed.2024.107537. Epub 2024 Jan 20. PMID 38253245
- [Derived] DeLeon S, Barsanti F, Holweg CTJ, Yoo B, Creasy B, Wechsler ME. Omalizumab treatment reduces asthma exacerbations regardless of airway bronchodilator reversibility. J Allergy Clin Immunol Pract. 2022 Aug;10(8):2181-2183.e1. doi: 10.1016/j.jaip.2022.04.029. Epub 2022 May 6. No abstract available. PMID 35526776
- [Derived] Soong W, Yoo B, Pazwash H, Holweg CTJ, Casale TB. Omalizumab response in patients with asthma by number and type of allergen. Ann Allergy Asthma Immunol. 2021 Aug;127(2):223-231. doi: 10.1016/j.anai.2021.04.002. Epub 2021 Apr 8. PMID 33838339
- [Derived] Chen M, Choo E, Yoo B, Raut P, Haselkorn T, Pazwash H, Holweg CTJ, Hudes G. No difference in omalizumab efficacy in patients with asthma by number of asthma-related and allergic comorbidities. Ann Allergy Asthma Immunol. 2021 Jun;126(6):666-673. doi: 10.1016/j.anai.2021.01.015. Epub 2021 Jan 17. PMID 33465457
- [Derived] Chen M, Shepard K 2nd, Yang M, Raut P, Pazwash H, Holweg CTJ, Choo E. Overlap of allergic, eosinophilic and type 2 inflammatory subtypes in moderate-to-severe asthma. Clin Exp Allergy. 2021 Apr;51(4):546-555. doi: 10.1111/cea.13790. Epub 2021 Jan 7. PMID 33217063
- [Derived] Hanania NA, Djukanovic R, Heaney LG, Yang M, Yoo B, Iqbal A, Griffin NM, Chipps BE. Determinants of lung function improvement with omalizumab in adults with allergic asthma. J Allergy Clin Immunol Pract. 2020 Jun;8(6):2068-2070. doi: 10.1016/j.jaip.2020.01.019. Epub 2020 Jan 22. No abstract available. PMID 31981731
- [Derived] Hanania NA, Chipps BE, Griffin NM, Yoo B, Iqbal A, Casale TB. Omalizumab effectiveness in asthma-COPD overlap: Post hoc analysis of PROSPERO. J Allergy Clin Immunol. 2019 Apr;143(4):1629-1633.e2. doi: 10.1016/j.jaci.2018.11.032. Epub 2018 Dec 18. No abstract available. PMID 30576755
- [Derived] Luskin AT, Chipps BE, Casale TB, Griffin NM. Baseline asthma burden, comorbidities, and biomarkers in omalizumab-treated patients in PROSPERO. Ann Allergy Asthma Immunol. 2018 May;120(5):549-550. doi: 10.1016/j.anai.2018.01.034. Epub 2018 Feb 5. No abstract available. PMID 29421314
- [Derived] Chipps BE, Zeiger RS, Luskin AT, Busse WW, Trzaskoma BL, Antonova EN, Pazwash H, Limb SL, Solari PG, Griffin NM, Casale TB. Baseline asthma burden, comorbidities, and biomarkers in omalizumab-treated patients in PROSPERO. Ann Allergy Asthma Immunol. 2017 Dec;119(6):524-532.e2. doi: 10.1016/j.anai.2017.09.056. Epub 2017 Oct 18. PMID 29054589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are reported by age group (adult participants and adolescent participants) as well as for all participants.
Groups:
- Participants With Allergic Asthma (Age 12-17 Years): Adolescent participants (age 12-17 years) with allergic asthma, who had decided to initiate treatment with omalizumab were observed until a maximum follow-up of 12 months, death, withdrawal of consent, loss to follow-up, or study closure, whichever occurred first.
- Participants With Allergic Asthma (Age >/=18 Years): Adult participants (age greater than or equal to [>/=18] years) with allergic asthma, who had decided to initiate treatment with omalizumab were observed until a maximum follow-up of 12 months, death, withdrawal of consent, loss to follow-up, or study closure, whichever occurred first.
Period: Overall Study
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years)
Started | 69 | 737
Treated | 69 | 732
Completed | 59 | 563
Not Completed | 10 | 174
Not completed — Withdrawal by Subject | 2 | 44
Not completed — Adverse Event | 1 | 7
Not completed — Death | 0 | 5
Not completed — Pregnancy | 0 | 2
Not completed — Participant non-compliance | 4 | 46
Not completed — Investigator/Sponsor decision | 1 | 4
Not completed — Other unspecified | 2 | 66

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Participants With Allergic Asthma (Age >/=18 Years): Adult participants (age >/=18 years) with allergic asthma, who had decided to initiate treatment with omalizumab were observed until a maximum follow-up of 12 months, death, withdrawal of consent, loss to follow-up, or study closure, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total
Number analyzed (Participants) | 69 | 737 | 806
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (1.69) | 50.4 (14.75) | 47.3 (17.40)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All enrolled participants
  Participants
    Female | 25 | 487 | 512
    Male | 44 | 250 | 294

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Asthma Exacerbations During Months 1-12
Description: An asthma exacerbation was defined as new or increased asthma symptoms which resulted in either hospitalization and/or treatment with systemic corticosteroids (or increase of stable maintenance dose) for >/= 3 days.
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma exacerbations
Groups:
- Total Participants With Allergic Asthma: All participants with allergic asthma, who had decided to initiate treatment with omalizumab were observed until a maximum follow-up of 12 months, death, withdrawal of consent, loss to follow-up, or study closure, whichever occurred first.
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
asthma exacerbations | 0.46 (0.815) | 0.81 (1.407) | 0.78 (1.369)

2. Secondary Outcome: Total Number of Asthma Exacerbations During Months 1-6
Description: An asthma exacerbation was defined as new or increased asthma symptoms which resulted in either hospitalization and/or treatment with systemic corticosteroids (or increase of stable maintenance dose) for >/=3 days.
Time Frame: Months 1-6
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma exacerbations
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 726 | 795
asthma exacerbations | 0.20 (0.440) | 0.51 (0.988) | 0.48 (0.957)

3. Secondary Outcome: Total Number of Asthma Exacerbations During Months 7-12
Description: as for outcome 1
Time Frame: Months 7-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma exacerbations
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 635 | 698
asthma exacerbations | 0.29 (0.521) | 0.35 (0.756) | 0.35 (0.738)

4. Secondary Outcome: Total Number of Asthma-Related Hospital Admissions During Months 1-12
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related hospital admissions
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
asthma-related hospital admissions | 0.04 (0.205) | 0.06 (0.356) | 0.06 (0.346)

5. Secondary Outcome: Total Number of Asthma-Related Hospital Admissions During Months 1-6
Time Frame: Months 1-6
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related hospital admissions
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 726 | 795
asthma-related hospital admissions | 0.03 (0.169) | 0.03 (0.230) | 0.03 (0.225)

6. Secondary Outcome: Total Number of Asthma-Related Hospital Admissions During Months 7-12
Time Frame: Months 7-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related hospital admissions
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 635 | 698
asthma-related hospital admissions | 0.02 (0.126) | 0.03 (0.215) | 0.03 (0.208)

7. Secondary Outcome: Total Number of Asthma-Related ER Visits During Months 1-12
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related ER visits
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
asthma-related ER visits | 0.13 (0.380) | 0.14 (0.575) | 0.14 (0.560)

8. Secondary Outcome: Total Number of Asthma-Related Emergency Room (ER) Visits During Months 1-6
Time Frame: Months 1-6
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related ER visits
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 726 | 795
asthma-related ER visits | 0.04 (0.205) | 0.09 (0.410) | 0.09 (0.397)

9. Secondary Outcome: Total Number of Asthma-Related ER Visits During Months 7-12
Time Frame: Months 7-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related ER visits
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 635 | 698
asthma-related ER visits | 0.10 (0.296) | 0.06 (0.293) | 0.06 (0.294)

10. Secondary Outcome: Total Number of Asthma-Related Unscheduled Physician's Office Visits During Months 1-12
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related physician's office visits
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
asthma-related physician's office visits | 0.39 (0.771) | 0.39 (0.866) | 0.39 (0.858)

11. Secondary Outcome: Total Number of Asthma-Related Unscheduled Physician's Office Visits During Months 1-6
Time Frame: Months 1-6
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related physician's office visits
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 726 | 795
asthma-related physician's office visits | 0.23 (0.598) | 0.23 (0.584) | 0.23 (0.585)

12. Secondary Outcome: Total Number of Asthma-Related Unscheduled Physician's Office Visits During Months 7-12
Time Frame: Months 7-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related physician's office visits
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 635 | 698
asthma-related physician's office visits | 0.17 (0.423) | 0.18 (0.515) | 0.18 (0.507)

13. Secondary Outcome: Total Number of Asthma-Related Telephone Calls to Healthcare Providers During Months 1-12
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related telephone calls
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
asthma-related telephone calls | 0.35 (0.783) | 0.43 (1.181) | 0.43 (1.152)

14. Secondary Outcome: Total Number of Asthma-Related Telephone Calls to Healthcare Providers During Months 1-6
Time Frame: Months 1-6
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related telephone calls
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 726 | 795
asthma-related telephone calls | 0.16 (0.407) | 0.24 (0.799) | 0.23 (0.773)

15. Secondary Outcome: Total Number of Asthma-Related Telephone Calls to Healthcare Providers During Months 7-12
Time Frame: Months 7-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: asthma-related telephone calls
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 635 | 698
asthma-related telephone calls | 0.21 (0.544) | 0.22 (0.692) | 0.22 (0.680)

16. Secondary Outcome: Percentage of Participants by Number of Asthma Exacerbations
Description: Percentage of participants by number of asthma exacerbations (0, 1, 2, 3, >/=4) was reported. An asthma exacerbation was defined as new or increased asthma symptoms which resulted in either hospitalization and/or treatment with systemic corticosteroids (or increase of stable maintenance dose) for >/= 3 days.
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
percentage of participants
  No (0) Asthma Exacerbation | 69.6 | 61.8 | 62.4
  1 Asthma Exacerbation | 18.8 | 18.3 | 18.3
  2 Asthma Exacerbations | 7.2 | 9.2 | 9.0
  3 Asthma Exacerbations | 4.3 | 4.3 | 4.3
  >/=4 Asthma Exacerbations | 0 | 6.5 | 5.9

17. Secondary Outcome: Percentage of Participants by Number of Asthma Exacerbations Requiring Treatment With Systemic Steroids
Description: Percentage of participants by number of asthma exacerbations (0, 1, 2, 3, >/=4) requiring treatment with systemic steroids was reported. An asthma exacerbation was defined as new or increased asthma symptoms which resulted in either hospitalization and/or treatment with systemic corticosteroids (or increase of stable maintenance dose) for >/= 3 days.
Time Frame: Months 1-12
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 727 | 796
percentage of participants
  No (0) Asthma Exacerbation Requiring Treatment | 71.0 | 62.3 | 63.1
  1 Asthma Exacerbation Requiring Treatment | 20.3 | 18.2 | 18.3
  2 Asthma Exacerbations Requiring Treatment | 4.3 | 9.4 | 8.9
  3 Asthma Exacerbations Requiring Treatment | 4.3 | 4.5 | 4.5
  >/=4 Asthma Exacerbations Requiring Treatment | 0 | 5.6 | 5.2

18. Secondary Outcome: Change From Baseline in Raw Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 was defined as the volume of air that can be forced out in one second after taking a deep breath. Pre-bronchodilator FEV1 and post-bronchodilator FEV1 are reported for each timepoint. FEV1 was measured using spirometry.
Time Frame: Baseline, Month 6, end of study (EOS)/early termination (ET) (up to Month 12)
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure. Here, number analyzed=participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 67 | 728 | 795
liters
  Baseline: Pre-bronchodilator FEV1 | 2.61 (0.736) | 2.24 (0.820) | 2.27 (0.819)
  Change at Month 6: Pre-bronchodilator FEV1: number analyzed (Participants) | 58 | 568 | 626
  Change at Month 6: Pre-bronchodilator FEV1 | 0.09 (0.402) | 0.06 (0.359) | 0.06 (0.363)
  Change at EOS/ET: Pre-bronchodilator FEV1: number analyzed (Participants) | 57 | 573 | 630
  Change at EOS/ET: Pre-bronchodilator FEV1 | 0.16 (0.463) | 0.03 (0.378) | 0.04 (0.388)
  Baseline: Post-bronchodilator FEV1: number analyzed (Participants) | 65 | 713 | 778
  Baseline: Post-bronchodilator FEV1 | 2.79 (0.767) | 2.38 (0.810) | 2.41 (0.814)
  Change at Month 6: Post-bronchodilator FEV1: number analyzed (Participants) | 54 | 523 | 577
  Change at Month 6: Post-bronchodilator FEV1 | 0.05 (0.522) | 0.04 (0.286) | 0.05 (0.315)
  Change at EOS/ET: Post-bronchodilator FEV1: number analyzed (Participants) | 52 | 534 | 586
  Change at EOS/ET: Post-bronchodilator FEV1 | 0.18 (0.446) | 0.02 (0.322) | 0.03 (0.338)

19. Secondary Outcome: Change From Baseline in Raw Forced Vital Capacity (FVC)
Description: FVC was defined as the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Pre-bronchodilator FVC and post-bronchodilator FVC are reported for each timepoint. FVC was measured using spirometry.
Time Frame: Baseline, Month 6, EOS/ET (up to Month 12)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 67 | 728 | 795
liters
  Baseline: Pre-bronchodilator FVC | 3.36 (0.842) | 3.08 (0.987) | 3.11 (0.978)
  Change at Month 6: Pre-bronchodilator FVC: number analyzed (Participants) | 57 | 568 | 625
  Change at Month 6: Pre-bronchodilator FVC | 0.09 (0.380) | 0.07 (0.562) | 0.07 (0.548)
  Change at EOS/ET: Pre-bronchodilator FVC: number analyzed (Participants) | 57 | 572 | 629
  Change at EOS/ET: Pre-bronchodilator FVC | 0.22 (0.321) | 0.03 (0.417) | 0.04 (0.413)
  Baseline: Post-bronchodilator FVC: number analyzed (Participants) | 65 | 713 | 778
  Baseline: Post-bronchodilator FVC | 3.43 (0.878) | 3.19 (0.959) | 3.21 (0.954)
  Change at Month 6: Post-bronchodilator FVC: number analyzed (Participants) | 53 | 523 | 576
  Change at Month 6: Post-bronchodilator FVC | 0.06 (0.324) | 0.07 (0.661) | 0.07 (0.637)
  Change at EOS/ET: Post-bronchodilator FVC: number analyzed (Participants) | 52 | 533 | 585
  Change at EOS/ET: Post-bronchodilator FVC | 0.20 (0.301) | 0.02 (0.349) | 0.04 (0.348)

20. Secondary Outcome: Change From Baseline in Raw Forced Expiratory Flow at 25-75 Percent (%) of Pulmonary Volume (FEF25%-75%)
Description: FEF25%-75% was defined as the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration. Pre-bronchodilator FEF25%-75% and post-bronchodilator FEF25%-75% are reported for each timepoint. FEF25%-75% was measured using spirometry.
Time Frame: Baseline, Month 6, EOS/ET (up to Month 12)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liters per second
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 67 | 727 | 794
liters per second
  Baseline:Pre-bronchodilator FEF25%-75% | 3.96 (12.328) | 2.28 (9.646) | 2.42 (9.902)
  Change at Month 6:Pre-bronchodilator FEF25%-75%: number analyzed (Participants) | 57 | 564 | 621
  Change at Month 6:Pre-bronchodilator FEF25%-75% | -1.66 (13.518) | -0.44 (10.868) | -0.55 (11.131)
  Change at EOS/ET:Pre-bronchodilator FEF25%-75%: number analyzed (Participants) | 57 | 568 | 625
  Change at EOS/ET:Pre-bronchodilator FEF25%-75% | -1.69 (13.426) | -0.47 (10.825) | -0.58 (11.080)
  Baseline:Post-bronchodilator FEF25%-75%: number analyzed (Participants) | 65 | 712 | 777
  Baseline:Post-bronchodilator FEF25%-75% | 3.76 (6.676) | 2.58 (9.503) | 2.68 (9.302)
  Change at Month 6:Post-bronchodilator FEF25%-75%: number analyzed (Participants) | 53 | 518 | 571
  Change at Month 6:Post-bronchodilator FEF25%-75% | -1.00 (7.513) | -0.59 (11.051) | -0.63 (10.767)
  Change at EOS/ET:Post-bronchodilator FEF25%-75%: number analyzed (Participants) | 52 | 530 | 582
  Change at EOS/ET:Post-bronchodilator FEF25%-75% | -0.76 (7.515) | -0.61 (10.926) | -0.62 (10.661)

21. Secondary Outcome: Change From Baseline in Percentage Predicted FEV1 (ppFEV1)
Description: FEV1 is the volume of air that can be forced out in one second after taking a deep breath, as measured using spirometry. Hankinson and Wang standards were used to calculate ppFEV1 (for age, gender, race, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. ppFEV1= 100 multiplied by (*) FEV1 (in liters [L]) divided by (/) predicted FEV1 (in L). Pre-bronchodilator ppFEV1 and post-bronchodilator ppFEV1 are reported for each timepoint.
Time Frame: Baseline, Month 6, EOS/ET (up to Month 12)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 67 | 728 | 795
percentage of predicted FEV1
  Baseline: Pre-bronchodilator ppFEV1 | 87.89 (16.934) | 74.23 (20.569) | 75.38 (20.631)
  Change at Month 6: Pre-bronchodilator ppFEV1: number analyzed (Participants) | 58 | 568 | 626
  Change at Month 6: Pre-bronchodilator ppFEV1 | 2.72 (13.279) | 1.77 (12.270) | 1.86 (12.359)
  Change at EOS/ET: Pre-bronchodilator ppFEV1: number analyzed (Participants) | 57 | 573 | 630
  Change at EOS/ET: Pre-bronchodilator ppFEV1 | 6.00 (14.713) | 0.91 (12.922) | 1.37 (13.163)
  Baseline: Post-bronchodilator ppFEV1: number analyzed (Participants) | 65 | 713 | 778
  Baseline: Post-bronchodilator ppFEV1 | 93.61 (16.416) | 78.92 (19.514) | 80.15 (19.690)
  Change at Month 6: Post-bronchodilator ppFEV1: number analyzed (Participants) | 54 | 523 | 577
  Change at Month 6: Post-bronchodilator ppFEV1 | 2.09 (16.398) | 1.47 (9.617) | 1.52 (10.421)
  Change at EOS/ET: Post-bronchodilator ppFEV1: number analyzed (Participants) | 52 | 534 | 586
  Change at EOS/ET: Post-bronchodilator ppFEV1 | 7.39 (14.673) | 0.82 (11.099) | 1.40 (11.597)

22. Secondary Outcome: Percentage of Participants With Prior Asthma Medications by Category or Class of Medications
Description: Prior asthma medications were defined as all medications used for asthma prior to the study (initiated within 90 days of baseline) and were assessed retrospectively at baseline. Participants received prior asthma medications of following categories or classes: short acting beta agonist (SABA), combination inhaled corticosteroids/long acting beta agonist (ICS/LABA), leukotriene receptor antagonist (LTRA), inhaled corticosteroids (ICS), oral/parenteral (systemic) corticosteroids, anticholinergic, long acting beta agonist (LABA), and other medication.
Time Frame: Baseline
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 737 | 806
percentage of participants
  All types | 98.6 | 99.3 | 99.3
  SABA | 91.3 | 88.6 | 88.8
  Combination ICS/LABA | 79.7 | 84.1 | 83.7
  LTRA | 73.9 | 66.6 | 67.2
  ICS | 36.2 | 33.8 | 34.0
  Oral/Parenteral (systemic) corticisteroids | 27.5 | 31.6 | 31.3
  Anticholinergic | 10.1 | 28.4 | 26.8
  LABA | 1.4 | 4.1 | 3.8
  Other medication | 5.8 | 5.3 | 5.3

23. Secondary Outcome: Percentage of Participants With Concomitant and Ongoing Asthma Medications by Category or Class of Medications
Description: Concomitant and ongoing asthma medications were defined as all medications used for asthma which began on or after the participant's study start, as well as those ongoing at the beginning of the study. Participants received following categories or classes of concomitant and ongoing asthma medications: SABA, combination ICS/LABA, LTRA, oral/parenteral (systemic) corticosteroids, ICS, anticholinergic, LABA, and other medication.
Time Frame: Baseline until EOS/ET (up to Month 12)
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 737 | 806
percentage of participants
  All types | 100.0 | 99.2 | 99.3
  SABA | 91.3 | 89.4 | 89.6
  Combination ICS/LABA | 82.6 | 82.4 | 82.4
  LTRA | 69.6 | 63.9 | 64.4
  Oral/Parenteral (systemic) corticosteroids | 37.7 | 47.2 | 46.4
  ICS | 33.3 | 34.3 | 34.2
  Anticholinergic | 11.6 | 32.6 | 30.8
  LABA | 1.4 | 4.5 | 4.2
  Other medication | 7.2 | 9.9 | 9.7

24. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ +12) Overall Score
Description: AQLQ +12 is a 32-item disease specific questionnaire designed to assess the participants' asthma-specific health-related quality of life (QOL). The questionnaire contains four domains: activity limitations (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). All items are scored on a 7-point likert scale. All item scores are averaged to produce one overall QOL score. Overall score ranges from 1 (total impairment) to 7 (no impairment), with higher scores indicating better QOL. A positive change from baseline indicated improved QOL.
Time Frame: Baseline, Month 6, EOS/ET (up to Month 12)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 69 | 732 | 801
units on a scale
  Baseline | 4.71 (1.332) | 3.93 (1.348) | 4.00 (1.363)
  Change at Month 6: number analyzed (Participants) | 59 | 593 | 652
  Change at Month 6 | 0.94 (1.134) | 1.18 (1.223) | 1.16 (1.216)
  Change at EOS/ET: number analyzed (Participants) | 63 | 603 | 666
  Change at EOS/ET | 1.11 (1.174) | 1.33 (1.267) | 1.31 (1.259)

25. Secondary Outcome: Change From Baseline in Asthma Control Test (ACT) Overall Score
Description: Multidimensional factors associated with asthma control from the participant's perspective were assessed using the ACT questionnaire. The ACT is a validated, five-item patient-reported outcome (PRO) questionnaire that measures the impact of asthma on home and work activities, shortness of breath, symptoms, rescue medication usage, and overall asthma control. All items are scored on a 5-point likert scale (1 to 5). All item scores are added together to calculate a total score. Total score ranges from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. A positive change from baseline indicated improvement.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 68 | 732 | 800
units on a scale
  Baseline | 16.40 (5.117) | 13.71 (4.910) | 13.94 (4.981)
  Change at Month 3: number analyzed (Participants) | 66 | 718 | 784
  Change at Month 3 | 3.11 (4.141) | 3.58 (4.263) | 3.54 (4.252)
  Change at Month 6: number analyzed (Participants) | 67 | 721 | 788
  Change at Month 6 | 3.57 (4.339) | 4.16 (4.677) | 4.11 (4.649)
  Change at Month 9: number analyzed (Participants) | 67 | 721 | 788
  Change at Month 9 | 3.90 (4.844) | 4.39 (4.910) | 4.35 (4.903)
  Change at Month 12: number analyzed (Participants) | 67 | 721 | 788
  Change at Month 12 | 3.90 (4.997) | 4.48 (4.926) | 4.43 (4.932)

26. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Asthma Questionnaire Score
Description: WPAI-asthma is a self-administered instrument to measure asthma-specific performance impairment of work and regular daily activity within the last 7 days and yields 4 types of scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (WI) (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). Total score and each score ranged from 0 (not affected/no impairment) to 100 (completely affected/impaired). Higher scores indicated greater impairment and less productivity. A negative change in score indicated improvement and a positive change indicated impairment.
Time Frame: Baseline, Month 6, EOS/ET (up to Month 12)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 67 | 717 | 784
units on a scale
  Work time missed: Baseline: number analyzed (Participants) | 3 | 401 | 404
  Work time missed: Baseline | 10.37 (14.759) | 7.70 (19.936) | 7.72 (19.890)
  Work time missed: Change at Month 6: number analyzed (Participants) | 1 | 297 | 298
  Work time missed: Change at Month 6 | 0.00 | -3.31 (19.796) | -3.30 (19.763)
  Work time missed: Change at EOS/ET: number analyzed (Participants) | 1 | 302 | 303
  Work time missed: Change at EOS/ET | -27.27 | -4.06 (21.977) | -4.14 (21.982)
  Impairment while working: Baseline: number analyzed (Participants) | 4 | 397 | 401
  Impairment while working: Baseline | 10.00 (14.142) | 31.36 (27.111) | 31.15 (27.087)
  Impairment while working: Change at Month 6: number analyzed (Participants) | 2 | 303 | 305
  Impairment while working: Change at Month 6 | 0.00 (0.000) | -16.24 (26.775) | -16.13 (26.719)
  Impairment while working: Change at EOS/ET: number analyzed (Participants) | 1 | 300 | 301
  Impairment while working: Change at EOS/ET | -30.00 | -15.93 (27.677) | -15.98 (27.643)
  Overall WI: Baseline: number analyzed (Participants) | 3 | 387 | 390
  Overall WI: Baseline | 20.85 (25.366) | 33.59 (28.737) | 33.49 (28.705)
  Overall WI: Change at Month 6: number analyzed (Participants) | 1 | 284 | 285
  Overall WI: Change at Month 6 | 0.00 | -15.55 (27.476) | -15.49 (27.443)
  Overall WI: Change at EOS/ET: number analyzed (Participants) | 1 | 286 | 287
  Overall WI: Change at EOS/ET | -49.09 | -16.24 (29.578) | -16.35 (29.590)
  Activity impairment: Baseline | 36.12 (27.577) | 48.79 (28.749) | 47.70 (28.893)
  Activity impairment: Change at Month 6: number analyzed (Participants) | 57 | 571 | 628
  Activity impairment: Change at Month 6 | -9.12 (33.449) | -19.30 (30.445) | -18.38 (30.840)
  Activity impairment: Change at EOS/ET: number analyzed (Participants) | 58 | 577 | 635
  Activity impairment: Change at EOS/ET | -14.83 (31.967) | -21.40 (32.424) | -20.80 (32.413)

27. Secondary Outcome: Percentage of Participants Who Showed an Improvement in Asthma Symptoms Due to the Medication, Assessed Using Global Evaluation of Treatment Effectiveness (GETE) by Inversigator
Description: Response to treatment was assessed using the GETE. The GETE is a validated instrument that measures the overall impression of the effect of the study medication on typical asthma symptoms. The evaluation was performed using the 5-point scale. The GETE scale ranges were as follows: 1=excellent, 2=good, 3=moderate, 4=poor, 5= worsening. A good or excellent response on the 5 point scale indicated that a participant had responded to treatment. Percentage of participants who showed an improvement (GETE scale score of 1 or 2) in asthma symptoms, as assessed by investigator, is reported.
Time Frame: EOS/ET (up to Month 12)
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 583 | 646
percentage of participants | 81.0 | 75.8 | 76.3

28. Secondary Outcome: Percentage of Participants Who Showed an Improvement in Asthma Symptoms Due to the Medication, Assessed Using GETE by Participant
Description: Response to treatment was assessed using the GETE. The GETE is a validated instrument that measures the overall impression of the effect of the study medication on typical asthma symptoms. The evaluation was performed using the 5-point scale. The GETE scale ranges were as follows: 1=excellent, 2=good, 3=moderate, 4=poor, 5= worsening. A good or excellent response on the 5 point scale indicated that a participant had responded to treatment. Percentage of participants who showed an improvement (GETE scale score of 1 or 2) in asthma symptoms, as assessed by participant, is reported.
Time Frame: EOS/ET (up to Month 12)
Population: All enrolled participants. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 63 | 599 | 662
percentage of participants | 87.3 | 75.0 | 76.1

29. Secondary Outcome: Change From Baseline in Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) Overall Quality of Life Score
Description: The MiniRQLQ is a shorter version of the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) instrument. The MiniRQLQ is a validated quality of life questionnaire to measure the functional impairments that are most troublesome to adult participants with either seasonal or perennial rhinoconjunctivitis of either allergic or non-allergic origin. The miniRQLQ contains 14 items; each item scored on a 7-point scale ranging from 0 [not impaired at all] to 6 [severely impaired]). The overall quality of life score is the average of the all item scores and ranges from 0 (not impaired at all) to 6 (severely impaired), with higher scores indicating more impairment. A negative change in score indicated improvement and a positive change indicated impairment.
Time Frame: Baseline, EOS/ET (up to Month 12)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Number analyzed (Participants) | 68 | 732 | 800
units on a scale
  Baseline | 2.44 (1.435) | 2.76 (1.375) | 2.73 (1.382)
  Change at EOS/ET: number analyzed (Participants) | 60 | 599 | 659
  Change at EOS/ET | -1.17 (1.357) | -0.99 (1.307) | -1.01 (1.311)

ADVERSE EVENTS:
Time Frame: From signing of informed consent form to 28 days after participants last visit (up to approximately 1 year)
Description: Safety evaluable participants defined as those who received at least 1 dose of omalizumab at any point in the study. Safety events collected and recorded during the study were: all serious adverse events, nonserious AEs of special interest, pregnancies, and nonserious AEs causally related to a Genentech product or where causality is unknown. Additional AEs not meeting the protocol-specified criteria listed above were reported during the study and were included in the safety database.
Arm/Group | Participants With Allergic Asthma (Age 12-17 Years) | Participants With Allergic Asthma (Age >/=18 Years) | Total Participants With Allergic Asthma
Serious Adverse Events (participants affected / at risk) | 5/69 | 85/732 | 90/801
Other Adverse Events (participants affected / at risk) | 9/69 | 58/732 | 67/801
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Allergic Asthma (Age 12-17 Years) (N=69) | Participants With Allergic Asthma (Age >/=18 Years) (N=732) | Total Participants With Allergic Asthma (N=801)
Acute left ventricular failure (Cardiac disorders) | 0 | 2 | 2
Myocardial infarction (Cardiac disorders) | 0 | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 2
Allergic granulomatous angiitis (Immune system disorders) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 11 | 11
Cellulitis (Infections and infestations) | 0 | 2 | 2
Diverticulitis (Infections and infestations) | 0 | 2 | 2
Influenza (Infections and infestations) | 1 | 1 | 2
Appendicitis (Infections and infestations) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Helicobacter test positive (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 2
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 23 | 26
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Mastectomy (Surgical and medical procedures) | 0 | 1 | 1
Muscle operation (Surgical and medical procedures) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Peripheral embolism (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Allergic Asthma (Age 12-17 Years) (N=69) | Participants With Allergic Asthma (Age >/=18 Years) (N=732) | Total Participants With Allergic Asthma (N=801)
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 2 | 2
Injection site reaction (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 1 | 1
Injection site pruritus (General disorders) | 0 | 1 | 1
Injection site swelling (General disorders) | 0 | 1 | 1
Local reaction (General disorders) | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Serum sickness (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 2
Acute sinusitis (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Mononucleosis syndrome (Infections and infestations) | 1 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Foot operation (Surgical and medical procedures) | 0 | 1 | 1
Hernia hiatus repair (Surgical and medical procedures) | 0 | 1 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 1
Meningioma surgery (Surgical and medical procedures) | 0 | 1 | 1
Rotator cuff repair (Surgical and medical procedures) | 0 | 1 | 1
Skin graft (Surgical and medical procedures) | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 3 | 3

LIMITATIONS AND CAVEATS:
This study was designed as an observational registry of participants with allergic asthma; but, was later reclassified as an interventional trial because the protocol was amended to include blood draws that were not considered to be standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.